CLINICAL TRIAL: NCT05854082
Title: How Related Are Speech Production and Reading? An Investigation of the Impact of Motor Tasks and Lidocaine on Reading Unfamiliar Words in Adults With and Without Dyslexia
Brief Title: Impact of Motor Tasks and Lidocaine on Reading Unfamiliar Words in Adults With and Without Dyslexia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00088290
Record Dates: First submitted 2023-03-28; First posted 2023-05-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Reading Disorders
MeSH Terms: conditions — Dyslexia | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Condition (Other): Typical Reader or Individual with Dyslexia
  Interventions: Drug: Lidocaine 2% Polyampoule

INTERVENTIONS:
Drug: Lidocaine 2% Polyampoule — Three intervention conditions in a repeated measures design - lidocaine; no perturbation, candy (lollipop)
  Other Names: No perturbation; Candy perturbation

SUMMARY:
Recent claims report that reading ability is partially dependent on speech production. While the evidence for this claim is compelling, it is not known to what extent, the speech production system contributes to successful reading performance in adult populations with dyslexia. One direct way to determine the influence of speech production feedback on reading performance is to measure reading performance in adults with dyslexia with an added motor component (i.e., sucking on a lollipop, holding a bite bar or numbing their oral mucosa with lidocaine).

To adults with and without dyslexia 18 years of age and older (60 in total; 30 in each group), three experimental tasks will be administered under four conditions (no motor task, lollipop, bite bar and lidocaine). The first task asks whether the letter string being presented is a word or a nonword. Secondly, a motor sequencing task will be administered where adults will be asked to label pictures. For all tasks, the accuracy and speed of responses will be measured by a computer while participants wear a fNIRS cap.

DETAILED DESCRIPTION:
While there are no clinical trials that have explored the explicit connection between reading and speech production (as the current study is proposing) the print-to-speech model provides a framework for understanding how the recognition of visual word forms (i.e., reading) is built upon acquisition and production of speech. Knowledge of how a word sounds and feels when produced (i.e., auditory and somatosensory feedback, respectively) scaffolds the development of knowledge about what a word looks like. This notion that reading development is heavily dependent on oral language skills follows from many studies providing evidence that oral language skills (i.e., vocabulary, syntax) and phonological awareness skills are predictors of both typical and deficient reading ability. Further, there are several nonclinical studies that provide convincing evidence that this connection needs to be better understood.

For example, children with apraxia of speech, a motor speech disorder that results in an impaired ability to plan and/or program the sequential movements required for speech that is not attributable to deficits in motor physiology (e.g., weakness, or spasticity) or deficits in language (i.e., reduced comprehension), are 1) at a high risk of developing a reading impairment and 2) have increased sensorimotor deficits. An investigation from 2009 evaluated the performance of 38 children with suspected apraxia of speech (CAS) on the Sensory Profile, a standardized assessment of sensory processing in children. Children with CAS had atypical sensory processing in five sensory factors, including oral sensory sensitivity. Increased oral sensory sensitivity in comparison to typically developing children has also been reported in children with specific language impairment, autism spectrum disorder (ASD) and attention deficit hyperactivity disorder (ADHD). In computational modelling, it has also been reported that the core impairment in CAS may be impaired feedforward commands secondary to reduced or degraded oral sensitivity, which fits well within the print-to-speech framework. An investigation of oral form discrimination performance in children with CAS (i.e., identification of geometric shapes in the mouth) reported that children with CAS scored significantly lower than typically developing children. Lower discrimination abilities are proposed to be an indicator of poor somatosensory function.

It has also been reported that sensory cueing approaches (which place emphasis on the relation between movements and auditory and somatosensory information via auditory, touch, pressure, kinesthetic and proprioceptive cues) are the most effective for treatment of CAS. Such results suggest that sensory cueing approaches either target the underlying impairment directly (i.e., restorative) or compensate for deficits (i.e., compensatory). The identification of sensory difficulties in children with CAS is important to understand speech characteristics and treatment efficacy in this population. These findings warrant additional investigations to understand if and to what extent somatosensory processing contributes to speech production and reading deficiencies in healthy and impaired adult and pediatric populations.

The investigators have found that oral form discrimination performance in adults is related to their reading performance and previously attempted to determine the influence of speech production feedback on reading performance by measuring reading performance in adults while adding an additional motor component (i.e., lollipop, bite bar, lidocaine). These somatosensory perturbations have the potential to alter and/or decrease the sensory feedback from the articulators in the mouth.

It was found that the lollipop had a facilitatory effect (i.e., faster response times) in the orthographic lexical decision tasks but no effect on the phonological lexical decision tasks or picture categorization tasks. In contrast, the lidocaine had a facilitatory effect (i.e., faster response times) in the phonological lexical decision tasks, but no facilitatory effects on the orthographic lexical decision tasks or picture categorization. Finally, the bite bar did not impact performance in any of the three tasks. However, it is not known if these effects (i.e., lollipop, bite bar, lidocaine) hold for an adult population with reading disorders. While completing these tasks under these conditions, brain activity will be measured using an functional near-infrared spectroscopy (fNIRS) system.

The approved investigational product is Lidocaine Hydrochloride Oral Topical Solution 2% USP. This oral topical anesthetic will temporarily numb the participant's articulators. This clinical trial will be conducted in compliance with this described protocol, good clinical practice (GCP) guidelines and the applicable regulatory requirement(s).

ELIGIBILITY:
Inclusion Criteria:

* All participants will be healthy and need to be proficient in English as the assessment materials are only available in English.
* Adult participants must weigh at least 50 kg or 110 lbs to avoid any possible toxic effects from the lidocaine.

Exclusion Criteria:

* Participants must have no personal or family history of adverse reactions to anesthetics to complete all the conditions.
* Participants who cannot consume sugary products will also be excluded.
* Additional exclusion criteria include: severe kidney disease; severe liver disease; treatment with class I antiarrhythmic drugs (such as mexiletine) or class III antiarrhythmic drugs (such as amiodarone)
* lack of integrity of oral mucosa]
* allergy to non-medicinal ingredients and preservatives (and related compounds) of Lidocaine Viscous, such as methylparaben, propylparaben, paraaminobenzoic acid, saccharin, artificial colours and flavour
* concomitant use of another anaesthetic containing lidocaine or another amide
* participant being pregnant or suspecting that she might be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Functional Near-InfraRed Spectroscopy (fNIRS) | 1 day
  Cortical activation in different brain regions using blood oxygenation changes measured using infrared light
Accuracy | 1 day
  Response to visually presented reading stimuli (i.e., correct or incorrect) recorded by the participant pressing on keyboard buttons
Response Time | 1 day
  Response time (in milliseconds) to visually presented reading stimuli recorded by the participant pressing on keyboard buttons

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Communication Sciences and Disorders, University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT05854082/Prot_SAP_001.pdf